CLINICAL TRIAL: NCT01403558
Title: Personality and Eating Behaviors in Morbidly Obese Patients
Acronym: PSYMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset i Vestfold HF (Other)
Collaborators: University of Tromso (Other)
Responsible Party: Principal Investigator, Hege Gade, PhD student, Sykehuset i Vestfold HF
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010/2071a
Record Dates: First submitted 2011-06-07; First posted 2011-07-27 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Eating Behaviors; Affective Symptoms
MeSH Terms: conditions — Feeding Behavior; Affective Symptoms | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive behavioral therapy (Experimental): Ten weekly individual cognitive behavioral therapy sessions before bariatric surgery
  Interventions: Behavioral: Cognitive behavioral therapy
- Control group (No Intervention): Usual preoperative care consisting of up to three voluntary sessions with nutritionist and physiotherapist before bariatric surgery

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — Cognitive behavioral therapy
  Arms: Cognitive behavioral therapy

SUMMARY:
The aim of this randomized controlled trial is assess the effect of a psychological based treatment model on eating behaviors and motivation for lifestyle changes in morbidly obese patients undergoing bariatric surgery.

Hypothesis: As compared with usual care, Cognitive Behavioral Therapy and Motivational interviewing-based (CBT/MI) intervention program will reduce dysfunctional eating behaviors and increase pre-surgical intrinsic motivation for lifestyle changes.

DETAILED DESCRIPTION:
Obesity is usually treated as a medical disease, prescribing interventions which adhere to the theoretically sound principles.The prevalence of obesity is increasing, and, accordingly, an increasing number of morbidly obese patients are eligible for Bariatric Surgery. This surgical procedure is highly effective and is often followed by resolution or remission of obesity related comorbidities (e.g. diabetes and obstructive sleep apnea). However, some individuals may have psychological and motivational problems that reduce these beneficial effects. Bariatric surgery represents a substantial part of total health care costs, and such costs may increase in the future. Another issue is that it is important to prevent post-surgical relapses. Hence, there is every reason to increase the effect and efficacy of both conservative treatments and bariatric surgery.

Clinically the investigators meet patients who regain their weight post-surgically, and the investigators have some experience that these patients may display more dysfunctional eating than those who are able to maintain a lower target weight. Given the expected outcome of the RCT, the autonomous motivation for lifestyle changes will be increased. Lowering dysfunctional eating, as well as increasing the probability of better success in preoperative weight loss, may help the patient to maintain a healthier weight after the surgical procedure. Moreover, developing a more tailored intervention for surgery patients may enable new evidence based treatments to be established for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been accepted for bariatric surgery

Exclusion Criteria:

* Patients suffering from drug and/or alcohol addiction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2011-09; Primary Completion 2020-03 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Change Eating behaviours | This co-primary outcome will be assessed, first, one week before the start of the 10 weeks intervention, and second, 1 week after the termination of the 10-weeks intervention. In addition a 1 and 4 year follow-up have been performed
  Eating behaviors: We will assess emotional eating, uncontrolled eating and Primary outcomes will be scored on the subscales "emotional eating" and "uncontrolled eating" on the TFEQ-R21. The predetermined criterion for clinically important improvement at 12 weeks will be a decrease of 15% from baseline on the emotional eating and uncontrolled eating subscale (range 0 to 100)
Change Affective symptoms | This co-primary outcome will be assessed, first, one week before the start of the 10 weeks intervention, and second, 1 week after the termination of the 10-weeks intervention. In addition a 1 and 4 year follow-up have been performed
  Affective symptoms will be assessed With the HADS

SECONDARY OUTCOMES:
Body weight - digital scale | As for primary outcome
  Body weight - digital scale (Soehnle Professional 2755)

OTHER OUTCOMES:
Health related quality of life - impact of weight on quality of life (IWQOL-lite) | 1 and 4 years after surgery
  Health related quality of life - impact of weight on quality of life (IWQOL-lite) is a 31-item questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jøran Hjelmesæth, PhD, Principal Investigator — Morbid Obesity Centre, Vestfold Hospital Trust, Tønsberg, Norway
Locations (2):
- Norway (2):
  - Hege Gade, Tønsberg, Vestfold
  - Senter for sykelig overvekt i Helse Sør-Øst, Sykehuset i Vestfold, Tønsberg

REFERENCES:
- [Derived] Hjelmesaeth J, Rosenvinge JH, Gade H, Friborg O. Effects of Cognitive Behavioral Therapy on Eating Behaviors, Affective Symptoms, and Weight Loss After Bariatric Surgery: a Randomized Clinical Trial. Obes Surg. 2019 Jan;29(1):61-69. doi: 10.1007/s11695-018-3471-x. PMID 30112603
- [Derived] Gade H, Friborg O, Rosenvinge JH, Smastuen MC, Hjelmesaeth J. The Impact of a Preoperative Cognitive Behavioural Therapy (CBT) on Dysfunctional Eating Behaviours, Affective Symptoms and Body Weight 1 Year after Bariatric Surgery: A Randomised Controlled Trial. Obes Surg. 2015 Nov;25(11):2112-9. doi: 10.1007/s11695-015-1673-z. PMID 25893651
- [Derived] Gade H, Hjelmesaeth J, Rosenvinge JH, Friborg O. Effectiveness of a cognitive behavioral therapy for dysfunctional eating among patients admitted for bariatric surgery: a randomized controlled trial. J Obes. 2014;2014:127936. doi: 10.1155/2014/127936. Epub 2014 Jul 21. PMID 25147733
- [Derived] Gade H, Rosenvinge JH, Hjelmesaeth J, Friborg O. Psychological correlates to dysfunctional eating patterns among morbidly obese patients accepted for bariatric surgery. Obes Facts. 2014;7(2):111-9. doi: 10.1159/000362257. Epub 2014 Mar 29. PMID 24685661